CLINICAL TRIAL: NCT00098371
Title: A Phase II Study of Flavopiridol Administered as a 30 Minute Loading Dose Followed by a 4-Hour Continuous Infusion in Patients With Previously Treated B-Cell Chronic Lymphocytic Leukemia or Prolymphocytic Leukemia Arising From CLL
Brief Title: Flavopiridol in Treating Patients With Chronic Lymphocytic Leukemia or Prolymphocytic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: CTEP Initiated Action.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00111; OSU 0491; N01CM62207 (NIH)
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-08

CONDITIONS: B-cell Chronic Lymphocytic Leukemia; Prolymphocytic Leukemia; Refractory Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic | interventions — alvocidib

ARMS (1):
- Treatment (alvocidib) (Experimental): Patients receive flavopiridol IV over 30 minutes followed by a 4-hour infusion on days 1, 8, 15, and 22. Treatment repeats every 42 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving at least a partial remission (PR) and whose PR lasts for > 6 months after completion of treatment may receive 6 additional courses of flavopiridol.
  Interventions: Drug: alvocidib

INTERVENTIONS:
Drug: alvocidib
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275

SUMMARY:
This phase II trial is studying how well flavopiridol works in treating patients with chronic lymphocytic leukemia or prolymphocytic leukemia. Drugs used in chemotherapy, such as flavopiridol, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the complete response (CR) and overall response rate (CR + Partial Response [PR]) of this regimen.

II. To assess the toxicity profile of this regimen. III. To examine response duration, progression-free survival and overall survival, following this treatment.

IV. To assess the pharmacokinetics of this novel schedule of administration.

SECONDARY OBJECTIVES:

I. To determine the influence of adverse prognostic factors including interphase cytogenetics, VH mutational status, ZAP-70 expression, CD38, and p53 mutational status with response to flavopiridol treatment.

II. To determine the influence of flavopiridol treatment on serial measurements of mcl-1 (mRNA and protein), HIF-1 (mRNA and protein), NF-kappaB activity, IkappaB, IkappaB phosphorylation, GSK-beta, and IL-6 down-stream targets.

III. To assess the relationship of drug induced apoptosis and mitochondrial perturbation of Chronic Lymphocytic Leukemia (CLL) cells in vitro and subsequent relationship to clinical response and tumor lysis in vivo.

IV. To examine cytokine levels (IL-6, IFN-gamma, TNF-alpha) during treatment with flavopiridol.

V. To assess pharmacokinetics (PK) to determine the variability of PK and PD analyses between treatment administrations and correlation with specific Single Nucleotide Polymorphisms (SNPs) potentially involved in flavopiridol disposition.

VI. To assess differences in diagnosis and relapse samples to investigate mechanisms of acquired flavopiridol resistance in primary CLL cells.

OUTLINE: This is an open-label study. Patients receive flavopiridol IV over 30 minutes followed by a 4-hour infusion on days 1, 8, 15, and 22.

Treatment repeats every 42 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving at least a partial remission (PR) and whose PR lasts for > 6 months after completion of treatment may receive 6 additional courses of flavopiridol.Patients are followed at 2 months and then every 3 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed B-cell chronic lymphocytic leukemia (CLL) or prolymphocytic leukemia (PLL) arising from CLL

  * No de novo PLL
  * Lymphocyte count > 5,000/mm^3 at some point since initial diagnosis of CLL
  * B-cells co-expressing CD5 AND CD19 or CD20
  * If no dim serum immunoglobulin or CD23 expression on leukemia cells, must be examined for cyclin D1 overexpression OR t(11;14) to rule out mantle cell lymphoma
* Requiring therapy, defined by any of the following:

  * Massive or progressive splenomegaly and/or lymphadenopathy
  * Anemia (hemoglobin < 11 g/dL) OR thrombocytopenia (platelet count < 100,000/mm^3)
  * Weight loss > 10% within the past 6 months
  * Grade 2 or 3 fatigue
  * Fevers > 100.5°C or night sweats for > 2 weeks with no evidence of infection
  * Progressive lymphocytosis with an increase of > 50% over a 2-month period OR an anticipated doubling time < 6 months
* Received ≥ 1 prior chemotherapy regimen that included fludarabine or nucleoside equivalent OR alternative therapy if contraindication to fludarabine exists (i.e., autoimmune hemolytic anemia)
* Performance status - ECOG 0-2
* More than 2 years
* See Disease Characteristics
* Baseline cytopenias allowed
* WBC ≤ 200,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN) (unless due to Gilbert's disease, hemolysis, or disease infiltration of the liver)
* AST ≤ 2 times ULN (unless due to hemolysis or disease infiltration of the liver)
* Creatinine ≤ 2.0 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy that would limit life expectancy
* See Disease Characteristics
* No other concurrent chemotherapy
* No concurrent chronic corticosteroids or corticosteroids as antiemetics
* No concurrent hormonal therapy except steroids for new adrenal failure or hormones for nondisease-related conditions (e.g., insulin for diabetes)
* No concurrent radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2005-04; Primary Completion 2009-06 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Byrd, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Result] Lin TS, Ruppert AS, Johnson AJ, Fischer B, Heerema NA, Andritsos LA, Blum KA, Flynn JM, Jones JA, Hu W, Moran ME, Mitchell SM, Smith LL, Wagner AJ, Raymond CA, Schaaf LJ, Phelps MA, Villalona-Calero MA, Grever MR, Byrd JC. Phase II study of flavopiridol in relapsed chronic lymphocytic leukemia demonstrating high response rates in genetically high-risk disease. J Clin Oncol. 2009 Dec 10;27(35):6012-8. doi: 10.1200/JCO.2009.22.6944. Epub 2009 Oct 13. PMID 19826119
- [Result] Pierceall WE, Warner SL, Lena RJ, Doykan C, Blake N, Elashoff M, Hoff DV, Bearss DJ, Cardone MH, Andritsos L, Byrd JC, Lanasa MC, Grever MR, Johnson AJ. Mitochondrial priming of chronic lymphocytic leukemia patients associates Bcl-xL dependence with alvocidib response. Leukemia. 2014 Nov;28(11):2251-4. doi: 10.1038/leu.2014.206. Epub 2014 Jul 3. No abstract available. PMID 24990615
- [Result] Woyach JA, Lozanski G, Ruppert AS, Lozanski A, Blum KA, Jones JA, Flynn JM, Johnson AJ, Grever MR, Heerema NA, Byrd JC. Outcome of patients with relapsed or refractory chronic lymphocytic leukemia treated with flavopiridol: impact of genetic features. Leukemia. 2012 Jun;26(6):1442-4. doi: 10.1038/leu.2011.375. Epub 2012 Jan 13. No abstract available. PMID 22289993
- [Derived] Yeh YY, Chen R, Hessler J, Mahoney E, Lehman AM, Heerema NA, Grever MR, Plunkett W, Byrd JC, Johnson AJ. Up-regulation of CDK9 kinase activity and Mcl-1 stability contributes to the acquired resistance to cyclin-dependent kinase inhibitors in leukemia. Oncotarget. 2015 Feb 20;6(5):2667-79. doi: 10.18632/oncotarget.2096. PMID 25596730

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Alvocidib): Patients receive flavopiridol IV over 30 minutes followed by a 4-hour infusion on days 1, 8, 15, and 22. Treatment repeats every 42 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving at least a partial remission (PR) and whose PR lasts for > 6 months after completion of treatment may receive 6 additional courses of flavopiridol.To improve tolerability of treatment regimen, an amendment to the protocol was done to reduce the cycle length from 42 days to 28 days, reducing the number of treatments per cycle from four (days 1, 8, 15 & 22) to three (days 1, 8, and 15).
Period: Overall Study
Arm/Group | Treatment (Alvocidib)
Started | 64
Completed | 64
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Alvocidib)
Number analyzed (Participants) | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 20
Age, Continuous [Median (Full Range); unit: years] | 60 [31 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 42
Region of Enrollment [Number; unit: participants]
  United States | 64

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate
Description: CR requires all of the following for at least two months from completion of therapy: Absence of lymphadenopathy in excess of 1 cm on physical exam; No hepatomegaly or splenomegaly on physical exam; Absence of constitutional symptoms; Normal CBC (complete blood count) as exhibited by polymorphonuclear leukocytes > 1500/µL, platelets > 100,000/µL, hemoglobin > 11.0 g/dl (untransfused); lymphocyte count < 5,000/µL; Bone marrow aspirate and biopsy must be normocellular for age with < 30% of nucleated cells being lymphocytes. Lymphoid nodules must be absent.
Time Frame: Up to 8 months
Population: Patients were assessed for clinical response after two, four and six cycles.
Measure: Number; unit: percent of patients
Arm/Group | Treatment (Alvocidib)
Number analyzed (Participants) | 64
percent of patients | 2

2. Primary Outcome: Overall Response Rate (CR + PR)
Description: CR requires all of the following: Absence of lymphadenopathy in excess of 1 cm on physical exam; No hepatomegaly or splenomegaly on physical exam; Absence of constitutional symptoms; Normal CBC as exhibited by polymorphonuclear leukocytes > 1500/µL, platelets > 100,000/µL, hemoglobin > 11.0 g/dl (untransfused); lymphocyte count < 5,000/µL; Bone marrow aspirate and biopsy must be normocellular for age with < 30% of nucleated cells being lymphocytes. Lymphoid nodules must be absent. Patients with CR after induction but wih treatment-related persistent cytopenia is a PR. PR requires a > 50% decrease in peripheral lymphocyte count from pretreatment value, > 50% reduction in lymphadenopathy, and/or > 50% reduction in splenomegaly/hepatomegaly. These patients must have one of the following: polymorphonuclear leukocytes > 1,500/μL , platelets > 100,000/μL, hemoglobin > 11.0 g/dl (untransfused) or any with 50% improvement from pretreatment value.
Time Frame: Up to 8 months
Population: Schedule was amended (cycle length) from 42 to 28 days, reduction in the number of doses per cycle from 4 to 3 and administration of prophylactic dexamethasone 20 mg IV on each treatment day.
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | Treatment (Alvocidib)
Number analyzed (Participants) | 64
percent of patients | 53 [41 to 65]

3. Primary Outcome: Response Duration
Description: Response evaluation criteria based on the Revised National Cancer Institute-sponsored Working Group Guidelines for response. Descriptive statistics will be computed (median, range, mean, standard deviation, minimum, and maximum) on response duration.
Time Frame: Up to 8 months
Population: Duration of response was not collected for patients.
Arm/Group | Treatment (Alvocidib)
Number analyzed (Participants) | 0

4. Primary Outcome: Progression-free Survival (PFS) for Responding Patients as Assessed Using Standard Kaplan-Meier Methods
Description: PFS was calculated from the date of study entry until time of disease progression or death, whichever came first, censoring patients alive and relapse free at last follow up. Patients who withdrew from study to undergo an allogeneic SCT (Stem cell transplantation) were censored at the time of transplantation.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Alvocidib)
Number analyzed (Participants) | 34
months | 12 [8.5 to 13.1]

5. Primary Outcome: Progression-free Survival for All Patients as Assessed Using Standard Kaplan-Meier Methods
Description: PFS was calculated from the date of study entry until time of disease progression or death, whichever came first, censoring patients alive and relapse free at last follow up. Patients who withdrew from study to undergo an allogeneic SCT were censored at the time of transplantation.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Alvocidib)
Number analyzed (Participants) | 64
months | 8.6 [6.7 to 12.6]

6. Primary Outcome: Overall Survival
Description: Overall survival data will be reported on a 3-month basis for 5 years
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Alvocidib)
Number analyzed (Participants) | 64
months | 28.8 [18.6 to 32.9]

7. Primary Outcome: Toxicity
Description: Toxicity determination based on NCI Common Toxicity Criteria version 3 and modified NCI Common toxicity guidelines for evaluating hematologic toxicity in leukemia.
Time Frame: Measurement prior to each infusion, at end of therapy, 2 months post-completion and post-treatment follow-up every 3 months for two years.
Population: Grade 3 to 4 infections requiring IV antibiotics and were generally related to upper or lower respiratory infections or infections of indwelling central venous catheters.
Measure: Number; unit: percentage of patients
Groups:
- Treatment (Alvocidib): Patients receive flavopiridol IV over 30 minutes followed by a 4-hour infusion on days 1, 8, 15, and 22. Treatment repeats every 42 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving at least a partial remission (PR) and whose PR lasts for > 6 months after completion of treatment may receive 6 additional courses of flavopiridol.
  alvocidib
Arm/Group | Treatment (Alvocidib)
Number analyzed (Participants) | 64
percentage of patients | 25

8. Secondary Outcome: Pharmacokinetics (PK) (AUC) as Assessed by Plasma Levels of Both Flavopiridol and Metabolites of Flavopiridol
Description: Pharmacokinetics were performed on day 1 and day 8 of cycle 1 by plasma levels of both flavopiridol and metabolites of flavopiridol using Area Under the Curve (AUC)
Time Frame: During treatment day 1 and day 8 of cycle 1
Population: The values are overall averages for all patients on days 1 and 8 - therefore, there is only a single value for each parameter.
Measure: Mean (Standard Deviation); unit: μM*hr
Arm/Group | Treatment (Alvocidib)
Number analyzed (Participants) | 63
μM*hr | 9.42 (5.11)

9. Secondary Outcome: PK (Cmax) as Assessed by Plasma Levels of Both Flavopiridol and Metabolites of Flavopiridol
Description: Pharmacokinetics were performed on day 1 and day 8 of cycle 1 by plasma levels of both flavopiridol and metabolites of flavopiridol
Time Frame: During treatment day 1 and day 8 of course 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: μM
Arm/Group | Treatment (Alvocidib)
Number analyzed (Participants) | 63
μM | 2.04 (1.05)

10. Secondary Outcome: PK as Assessed by Levels of Both Flavopiridol and Metabolites of Flavopiridol in Urine Samples
Description: urine samples were collected in some patients during the first 24 hours after the start of the infusion on cycle 1, day 1 to isolate metabolites of flavopiridol to be used as internal standard for plasma metabolite quantification experiments.
Time Frame: Urine collected at 4 separate times in some patients during the first 24 hours after start of infusion on day 1 of course 1.
Population: Data for this PK analysis was not collected and analyzed.
Arm/Group | Treatment (Alvocidib)
Number analyzed (Participants) | 0

11. Secondary Outcome: Serial Levels of IL-6 as Assessed by Blood Plasma
Description: IL-6 measures were adjusted for baseline values
Time Frame: 4.5 hours, 8 hours, 12 hours, and 24 hours following the initiation of therapy during day 1 of course 1
Population: IL-6 expression analysis was available for only day 1 and not day 8.
Measure: Mean (95% Confidence Interval); unit: pg/ml
Groups:
- Group 1: Patients without dexamethasone
- Group 2: Patients with dexamethasone
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 26 | 31
pg/ml
  4.5 hours | 3.5 [2.7 to 4.6] | 1.6 [1.2 to 2.0]
  8 hours | 13.4 [9.8 to 18.4] | 2.2 [1.7 to 2.9]
  12 hours | 25.5 [17.3 to 37.6] | 2.5 [1.8 to 3.6]
  24 hours | 13.2 [8.0 to 21.7] | 3.9 [2.5 to 6.2]

12. Secondary Outcome: Comparison of CLL Cell Samples Taken at Registration/Diagnosis to CLL Cell Samples Taken at Time of Relapse
Description: Samples will be examined for ex vivo sensitivity to flavopiridol, expression of select anti-apoptosis proteins, BCRP mRNA and protein expression, difference in gene expression by cDNA microarray and potentially by epigenetic arrays. Comparisons will be used to evaluate mechanisms of acquired flavopiridol resistance.
Time Frame: At baseline and at time of relapse or when patient goes off therapy due to disease progression
Population: Data for this outcome as not collected and analyzed
Arm/Group | Treatment (Alvocidib)
Number analyzed (Participants) | 0

13. Secondary Outcome: Correlation of Adverse Prognostic Factors With Response to Flavopiridol Treatment as Assessed by Interphase Cytogenetics, VH Mutational Status, ZAP-70 Protein Expression, CD38, and p53
Description: overall response rates (CR+PR)
Time Frame: up to 8 months
Population: Data were not collected and analyzed for VH mutational status, ZAP-70 protein expression, CD38, and p53
Measure: Number; unit: percentage of patients in each subgroup
Groups:
- Patients With Complex Karyotype: Complex Karyotype defined as three or more cytogenetic aberrations.
- Patients Without Complex Karyotype: Complex Karyotype defined as fewer than three cytogenetic aberrations.
Arm/Group | Patients With Del(17p13.1) | Patients Without Del(17p13.1) | Patients With Del(11q22.3) | Patients Without Del(11q22.3) | Patients With Complex Karyotype | Patients Without Complex Karyotype
Number analyzed (Participants) | 21 | 43 | 28 | 36 | 27 | 37
percentage of patients in each subgroup | 57 | 51 | 50 | 56 | 48 | 57

14. Secondary Outcome: Levels of Mcl-1 mRNA, Mcl-1 Protein, HIF-1alpha Protein, HIF-1alpha mRNA, NF-kappaB Activation, Total IkB, IkB Phosphorylation, GSK-beta Activity, and IL-6 Target Genes (i.e., STAT3)
Description: Assessed by real time RT-PCR (mcl-1, HIF-1alpha), immunoblot analysis (mcl-1, HIF-1alpha, I-kappaB, I-kappaB phosphorylation, targets of IL-6), and electrophoretic mobility shift analysis (NF-kappaB activation)
Time Frame: At baseline, 4.5 hours (end of continuous infusion), 8 hours, and approximately 24 hours following initiation of therapy
Population: Data was not collected and analyzed for this outcome
Arm/Group | Treatment (Alvocidib)
Number analyzed (Participants) | 0

15. Secondary Outcome: Comparison of Clinical Response and Tumor Lysis in Vivo With Drug-induced Apoptosis and Mitochondrial Perturbation in Vitro as Assessed by Flow Cytometry
Description: CLL cells will be incubated with control or flavopiridol (1 or 2.8 microMolar) for 4-hours followed by a 20 hours in media with 10% heat-inactivated human serum. Assessment of apoptosis following exposure of human CLL cells will be performed using annexin/PI flow cytometry. Patient samples with greater than 50% live cells (annexin-/PI-) following exposure to 2.8 microMolar flavopiridol will be considered to have insensitive disease. Patients whose CLL cells have less than 50% live cells at 1 microMolar will be considered to have highly sensitive disease.
Time Frame: At baseline
Population: A subset of patients who had sufficient material were analyzed according to response only.
Measure: Mean (Standard Deviation); unit: percentage of priming cells
Groups:
- Responders: Patients who achieved a partial response (PR)
- Non-Responders: Patients who had stable disease (SD) or progressive disease (PD)
Arm/Group | Responders | Non-Responders
Number analyzed (Participants) | 9 | 4
percentage of priming cells | 22.2 (16.5) | 6.4 (4.3)

ADVERSE EVENTS:
Description: NCI Common Toxicity Criteria of Adverse Events (version 3) and modified NCI Common Toxicity Criteria guidelines for evaluating hematologic toxicity for leukemia was used to grade adverse events for patients. Adverse events are reported across all grades.
Arm/Group | Treatment (Alvocidib)
Serious Adverse Events (participants affected / at risk) | 4/64
Other Adverse Events (participants affected / at risk) | 64/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Alvocidib) (N=64)
Infection (Infections and infestations) | 4 (4) — Serious Adverse events reported were deaths
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Alvocidib) (N=64)
Neutropenia (Investigations) | 62 (62)
Anemia (Blood and lymphatic system disorders) | 38 (38)
Thrombocytopenia (Injury, poisoning and procedural complications) | 42 (42)
Fatigue (General disorders) | 60 (60)
Diarrhea (Gastrointestinal disorders) | 60 (60)
Nausea and Vomiting (Gastrointestinal disorders) | 48 (48)
Anorexia (Metabolism and nutrition disorders) | 20 (20)
Anxiety/Depression (Psychiatric disorders) | 11 (11)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 28 (28)
Cytokine Release Syndrome (Immune system disorders) | 27 (27)
Transaminitis (Investigations) | 59 (59)
Hyperbilirubinemia (Investigations) | 15 (15)
Infection (Infections and infestations) | 43 (43)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less